CLINICAL TRIAL: NCT00116506
Title: A Phase II Study of Bevacizumab (Avastin™) and Erlotinib (Tarceva™) in Combination With FOLFOX for Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Study of Bevacizumab, Erlotinib, FOLFOX for Patients With Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry); Sanofi-Synthelabo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-365
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: Metastatic Colorectal Cancer; Bevacizumab; Erlotinib; FOLFOX
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Erlotinib Hydrochloride; Folfox protocol; Bevacizumab

INTERVENTIONS:
Drug: erlotinib
Drug: FOLFOX
Drug: bevacizumab

SUMMARY:
Despite recent advances, most patients with advanced colorectal cancer continue to have a poor prognosis. 5-FU, leucovorin, oxaliplatin and bevacizumab is a standard treatment option for patients with stage IV colorectal cancer. Fluorouracil (5-FU), leucovorin and oxaliplatin are considered traditional chemotherapies that try to stop tumor growth by affecting how they divide. Bevacizumab is a therapy to try to block the blood vessels that tumors need to grow. It is considered a 'targeted agent'. Erlotinib is another targeted agent, that has been shown to be effective in treating lung and other cancers. This trial is assessing the potential benefit of adding these second targeted agents to standard treatment.

DETAILED DESCRIPTION:
* Patients receive bevacizumab, oxaliplatin, leucovorin, and 5-FU intravenously. The erlotinib is taken orally each day. One cycle of study therapy is 14 days. Cycles may be repeated unless there are intolerable side effects or the cancer worsens.
* Patients will undergo a tumor measurement evaluation following 3 cycles of study therapy, and then every 4 cycles thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have histologically or cytologically documented locally advanced or metastatic colorectal cancer
* No prior chemotherapy treatment for advanced or metastatic colorectal cancer. Patients may have received prior adjuvant chemotherapy or radiation with radiosensitizing chemotherapy. The last course of adjuvant chemotherapy must have concluded > 12 months prior to registration. Patients may not have previously received irinotecan, oxaliplatin, antiangiogenesis agent, or EGFR inhibitor therapy in either the adjuvant or metastatic setting. No concurrent use of additional investigational agents (including up to 4 weeks prior to enrollment) is allowed while participating in this study.
* Palliative radiation for metastatic disease is allowed, however at least 4 weeks must elapse from last treatment to first cycle of therapy and patient must have fully recovered from side effects of radiation therapy.
* Patients must have measurable disease
* Age > 18 years.
* ECOG Performance Score of 0-1.
* Patients should have completed any major surgery > 4 weeks from registration. Patients must have completed any minor surgery (including CT or U/S guided biopsies) > 7 days from registration. Patients must have fully recovered from the procedure. (Insertion of a vascular access device is not considered major or minor surgery).
* Adequate bone marrow as evidenced by: *Absolute neutrophil count > 1,500/mL; *Platelet count > 100,000/mL
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL
* Adequate hepatic function as evidenced by: *Serum total bilirubin < 1.5 mg/dL; *Alkaline phosphatase < 3X the ULN (< 5X the ULN for patients with known hepatic metastases);

  * SGOT/SGPT < 3X the ULN (< 5X the ULN for patients with known hepatic metastases)
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication.

Exclusion Criteria:

* Patients with an active infection or with a fever within 3 days of the first scheduled day of protocol treatment.
* Presence of central nervous system or brain metastases.
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or treated localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry.
* Patients with known hypersensitivity to any of the components of oxaliplatin, 5-fluorouracil (or other fluoropyrimidines), leucovorin, bevacizumab or erlotinib.
* Peripheral neuropathy > Grade 2.
* Patients who are pregnant or lactating.
* Any other medical condition, including mental illness or substance abuse, deemed by the clinician to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant.
* Known HIV or Hepatitis B or C
* Inadequately controlled hypertension
* Unstable angina or New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction within 6 months.
* History of stroke within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Urine protein:creatinine ratio ≥ 1.0 at screening.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* Serious, non-healing wound, ulcer, or bone fracture.
* Patients lacking physical integrity of the upper gastrointestinal tract or who have malabsorption syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate 1 year progression-free survival

SECONDARY OUTCOMES:
Determination of the observed response rate, median duration of response and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusett General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts